CLINICAL TRIAL: NCT03541434
Title: Analysis of Clinical, Pathologic and Molecular Markers of Adenotonsillar Hypertrophic Disease
Brief Title: Bioclinical Profile of Adenotonsillar Hypertrophy in the Pediatric Population
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Georgios Stathopoulos, Associate Professor of Physiology, University of Patras
Other Study IDs: 14/30-09-2016 CHPatras
Record Dates: First submitted 2018-05-09; First posted 2018-05-30 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Enlargement of Tonsil or Adenoid
Keywords: obstructive sleep apnea; tonsillitis; middle ear effusion; pathophysiology; score
MeSH Terms: conditions — Sleep Apnea, Obstructive; Tonsillitis; Otitis Media with Effusion | interventions — Blood Cell Count; Acoustic Impedance Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood was centrifuged and cells were separated from supernatants. Both were stored at -80 degrees.
  Palatine and pharyngeal tonsillar tissue specimens were divided in half. One part was fixated in 4% formaldehyde for 24 hours and then stored in saline at 4 degrees. The other part was stored immediately at -80 degrees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy: Children with no history of adenotonsillar hypertrophy, recurrent tonsillitis, or middle ear effusion. They presented to the clinic for examination or a scheduled procedure.
  Interventions: Diagnostic Test: Complete Blood Count; Diagnostic Test: Tympanometry
- Recurrent tonsillitis: Children with a history of recurret tonsillitis but no adenotonsillar hypertrophy. Diagnosis was based on physical exam and complete blood count. They presented to the clinic for a sceduled tonsillectomy.
  Interventions: Diagnostic Test: Complete Blood Count; Diagnostic Test: Tympanometry; Procedure: Tonsillectomy and/or adenoidectomy
- Middle ear effusion: Children with chronic middle ear effusion but no adenotonsillar hypertrophy. Diagnosis was based on physical exam and tympanometry. They presented to the clinic for scheduled myringotomy with or without adenoidectomy.
  Interventions: Diagnostic Test: Complete Blood Count; Diagnostic Test: Tympanometry; Procedure: Tonsillectomy and/or adenoidectomy
- Adenotonsillar hypertrophy: Children with tonsillar and/or adenoidal hypertrophy. Diagnosis was based on physical exam and partly on x-ray of nasopharynx or nasopharyngoscopy. They presented to the clinic for scheduled tonsillectomy and/or adenoidectomy.
  Interventions: Diagnostic Test: Complete Blood Count; Diagnostic Test: Tympanometry; Procedure: Tonsillectomy and/or adenoidectomy

INTERVENTIONS:
Diagnostic Test: Complete Blood Count — White blood cell subgroups count
Diagnostic Test: Tympanometry — Conventional and multifrequency tympanometry, documenting middle ear admittance and absorbance
Procedure: Tonsillectomy and/or adenoidectomy — Excision of palatine and/or pharyngeal tonsils.
  Groups: Adenotonsillar hypertrophy; Middle ear effusion; Recurrent tonsillitis

SUMMARY:
Adenotonsillar hypertrophy is the principal cause of obstructive sleep apnea of childhood, yet little is known with regard to its pathophysiologic and molecular mechanisms. The present trial examines potential bioclinical markers of the disease.

DETAILED DESCRIPTION:
Background: Tonsils and adenoids comprise the main bulk of Waldeyer's ring, which is commonly enlarged in childhood, until the age of 11. Obstructive sleep apnea caused by adenotonsillar hypertrophy is a major contributing factor to cardiorespiratory morbidity in the pediatric population. It is also responsible for otitis media with effusion, the most frequent cause of children's hearing loss. Even so, there is scarce knowledge of its molecular pathogenesis.

Objective: Identification of clinical/molecular markers of adenotonsillar enlargement and investigation of their participation in the process of tissue hypertrophy.

Methods: A prospective cohort of children with adenotonsillar hypertrophy were recruited starting on 02/01/2017 and ending on 12/22/2017. Demographic and clinical data including age, gender, sleep apnea severity, tonsillar size, presence of middle ear effusion, family history, review of systems as well as tympanometric and complete blood count results were recorded. Blood samples and tissue specimens from the therapeutic adenotonsillectomy procedure were archived for future analyses. Children with chronic tonsillitis and/or adenoiditis, who also underwent excision of tonsils and/or adenoids served as study controls. Informed consent was obtained from parents of all study participants.

ELIGIBILITY:
Inclusion Criteria:

* Available history and physical exam findings
* Available complete blood count and tympanometry at admission

Exclusion Criteria:

* Previous tonsillectomy and/or adenoidectomy.
* Previous ear surgery.
* Acute infection during the past month.
* Active severe systemic disease.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children presenting to the clinics of a Pediatric hospital.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Bioclinical profile of adenotonsillar hypertrophy | One year post surgical procedure
  Clinical, laboratory, and molecular markers of adenotonsillar hypertrophy

SECONDARY OUTCOMES:
Clinical markers of adenotonsillar hypertrophy | One year post surgical procedure
  Clinical findings from history (sympoms) and physical exam (signs) suggestive of adenotonsillar hypertrophy.
Laboratory markers of adenotonsillar hypertrophy | One year post surgical procedure
  Complete blood count (cells/L)
Tympanometric findings of middle ear disease resulting from adenotonsillar hypertrophy | One year post surgical procedure
  Middle ear pressure (dekaPascals)
Wide-Band tympanometric findings of middle ear disease resulting from adenotonsillar hypertrophy | One year post surgical procedure
  Resonance frequency of the middle ear (Hz)
Molecular determinants of adenotonsillar hypertrophy | One year post surgical procedure
  Immunohistochemical expression of molecular factors involved in tissue growth (semiquantitative scale)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios T Stathopoulos, Principal Investigator — Associate Professor of Physiology
Locations (2):
- Greece (2):
  - Children Hospital of Patras "Karamandaneio", Pátrai, Achaia
  - Patras University Hospital, Rio, Achaia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Ward SD, Sheldon SH, Shiffman RN, Lehmann C, Spruyt K; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):e714-55. doi: 10.1542/peds.2012-1672. Epub 2012 Aug 27. PMID 22926176
- [Result] Liou HC. Regulation of the immune system by NF-kappaB and IkappaB. J Biochem Mol Biol. 2002 Nov 30;35(6):537-46. doi: 10.5483/bmbrep.2002.35.6.537. PMID 12470586
- [Result] Heneghan AF, Pierre JF, Kudsk KA. JAK-STAT and intestinal mucosal immunology. JAKSTAT. 2013 Oct 1;2(4):e25530. doi: 10.4161/jkst.25530. Epub 2013 Jun 26. PMID 24416649
- [Result] Min HJ, Kim SJ, Kim TH, Chung HJ, Yoon JH, Kim CH. Level of secreted HMGB1 correlates with severity of inflammation in chronic rhinosinusitis. Laryngoscope. 2015 Jul;125(7):E225-30. doi: 10.1002/lary.25172. Epub 2015 Jan 30. PMID 25639490
- [Derived] Kourelis K, Marazioti A, Kourelis T, Stathopoulos GT. Haematologic Markers and Tonsil-to-Body Weight Ratio to Assist Adenotonsillar Hypertrophy Diagnosis. Indian J Otolaryngol Head Neck Surg. 2022 Dec;74(Suppl 3):5604-5610. doi: 10.1007/s12070-021-02943-9. Epub 2021 Oct 25. PMID 36742935